CLINICAL TRIAL: NCT00287989
Title: A Randomized Phase II Trial Comparing Two Doses of Pulsed Erlotinib Prechemotherapy (PEP-C) in Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Brief Title: Erlotinib, Paclitaxel, and Carboplatin in Treating Patients With Stage III, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: J0432; P30CA006973 (NIH); JHOC-J0432; JHOC-WIRB-20041142; CDR0000455116 (Other: other); 20-04-11-42 (Other: JHM IRB)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Erlotinib Hydrochloride; Paclitaxel

ARMS (3):
- 150 PRE (Experimental): Erlotinib 150mg on days 1 and 2 of a 21 day cycle and Carboplatin AUC6 and Paclitaxel 200 mg/m2
  Interventions: Drug: Carboplatin; Drug: erlotinib hydrochloride; Drug: Paclitaxel
- 1,500 PRE (Experimental): Erlotinib 1500mg on Days 1 and 2 of a 21 day cycle and Carboplatin AUC6 and Paclitaxel 200mg/m2
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: erlotinib hydrochloride
- 1,500 POST (Experimental): Carboplatin AUC6, Paclitaxel 200 mg/m2 followed by Erlotinib 1500mg days 2 and 3.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: Carboplatin
  Other Names: Carboplatin AUC6
Drug: erlotinib hydrochloride — 150mg
  Other Names: Erlotinib
  Arms: 150 PRE
Drug: Paclitaxel — 200mg/m2
Drug: erlotinib hydrochloride — 1500mg
  Other Names: Erlotinib
  Arms: 1,500 POST; 1,500 PRE

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving erlotinib together with paclitaxel and carboplatin may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying two different doses of erlotinib when given together with paclitaxel and carboplatin to compare how well they work in treating patients with stage III, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the major objective response (complete and partial response) rates in patients with stage IIIB or IV or recurrent non-small cell lung cancer treated with high- versus low-dose erlotinib hydrochloride combined with paclitaxel and carboplatin.
* Compare the duration of response, time to progression, and survival of patients treated with these regimens.
* Characterize and compare the toxicities of these regimens.
* Determine the recommended phase III dose of erlotinib hydrochloride.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to gender. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral high-dose erlotinib hydrochloride on days 1 and 2. Patients also receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 3.
* Arm II: Patients receive oral low-dose erlotinib hydrochloride, paclitaxel, and carboplatin as in arm I.

In both arms, treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 58 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed non-small cell lung cancer

  * Stage IIIB or IV or recurrent disease
* Measurable or evaluable indicator lesions
* Must have smoked ≥ 100 cigarettes in his/her lifetime

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* WBC ≥ 4,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Bilirubin ≤ 1.0 mg/dL
* AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 week after completion of study treatment
* No gastrointestinal tract disease or inability to take oral medication
* No prior malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other active medical problems, including severe infection, unstable angina, or myocardial infarction within the past 6 months
* No poorly controlled hypertension or severe malnutrition
* No New York Heart Association class III or IV congestive heart failure or serious cardiac arrhythmia requiring medication except chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia)

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior radiotherapy to major bone marrow-containing sites
* No prior chemotherapy for advanced non-small cell lung cancer
* No prior agents directed at the epidermal growth factor receptor (EGFR)/HER axis (e.g., gefitinib, cetuximab, or trastuzumab [Herceptin®])
* No prior surgical procedure resulting in abnormal absorption of oral medications
* No concurrent surgical resection, palliative radiotherapy, or hormonal therapy
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-11; Primary Completion 2007-08 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Rudin, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Riely GJ, Rizvi NA, Kris MG, Milton DT, Solit DB, Rosen N, Senturk E, Azzoli CG, Brahmer JR, Sirotnak FM, Seshan VE, Fogle M, Ginsberg M, Miller VA, Rudin CM. Randomized phase II study of pulse erlotinib before or after carboplatin and paclitaxel in current or former smokers with advanced non-small-cell lung cancer. J Clin Oncol. 2009 Jan 10;27(2):264-70. doi: 10.1200/JCO.2008.17.4656. Epub 2008 Dec 1. PMID 19047285

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 150 PRE | 1,500 PRE | 1,500 POST
Started | 28 | 29 | 29
Completed | 28 | 29 | 29
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 PRE | 1,500 PRE | 1,500 POST | Total
Number analyzed (Participants) | 28 | 29 | 29 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 42
  >=65 years | 14 | 15 | 15 | 44
Age, Continuous [Median (Full Range); unit: years] | 68 [51 to 81] | 62 [42 to 78] | 62 [43 to 81] | 64 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 15 | 43
  Male | 13 | 16 | 14 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 29 | 29 | 86

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Percentage of patients who experienced complete or partial response as defined by RECIST
Time Frame: after 6 cycles of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 150 PRE | 1,500 PRE | 1,500 POST
Number analyzed (Participants) | 26 | 29 | 29
percentage of participants | 18 [6 to 37] | 34 [18 to 54] | 28 [13 to 47]

2. Secondary Outcome: Time to Progression
Description: Median number of months until disease progression
Time Frame: after cycle 6 of chemotherapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 150 PRE | 1,500 PRE | 1,500 POST
Number analyzed (Participants) | 28 | 29 | 29
months | 4 [3 to 5] | 4 [3 to 6] | 5 [3 to 8]

ADVERSE EVENTS:
Arm/Group | 150 PRE | 1,500 PRE | 1,500 POST
Serious Adverse Events (participants affected / at risk) | 5/28 | 9/29 | 8/29
Other Adverse Events (participants affected / at risk) | 2/28 | 2/29 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 PRE (N=28) | 1,500 PRE (N=29) | 1,500 POST (N=29)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 9 (9) | 8 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 PRE (N=28) | 1,500 PRE (N=29) | 1,500 POST (N=29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The design of the study was change during the course of this research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No